CLINICAL TRIAL: NCT02252653
Title: DISCOVERY: A Study Examining the Prevalence of TTR Mutations in Subjects Suspected of Having Cardiac Amyloidosis
Status: Completed | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-TTR-NT-002
Record Dates: First submitted 2014-09-22; First posted 2014-09-30 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Familial Amyloidotic Cardiomyopathy (FAC)
Keywords: Cardiomyopathy; Heart Failure; FAC; Amyloid; Transthyretin (TTR)
MeSH Terms: conditions — Cardiomyopathies; Heart Failure; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for TTR sequencing and cardiac function biomarkers; abdominal fat-pad aspirate for amyloid presence (optional for TTR positive patients only)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Familial Amyloidotic Cardiomyopathy (FAC)

SUMMARY:
The purpose of this study is to characterize the frequency of TTR mutations in subjects suspected of having cardiac amyloidosis

ELIGIBILITY:
Inclusion Criteria:

* Males or females >18 years old
* History of evidence suggestive of cardiac amyloidosis
* Subject is willing and able to comply with protocol required assessments and provide written informed consent

Exclusion Criteria:

* Known diagnosis of primary (AL) amyloidosis
* Known diagnosis of hereditary cardiomyopathy or cardiomyopathy due to aortic stenosis
* Patient is currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects Suspected of Having Familial Amyloidotic Cardiomyopathy (FAC)
Sampling Method: Non-Probability Sample
Enrollment: 1010 (Actual)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with of Transthyretin (TTR) mutations | Baseline
  Blood will be sequenced for the presence of TTR gene mutations

SECONDARY OUTCOMES:
Assessment of the presence of amyloid in tissue | Day 30
  An optional fine-needle aspirate of the abdominal fat pad will be collected
Quantification of biomarkers of cardiac function in serum | Day 30
  Biomarkers that assess cardiac function will be quantified from serum
Measurement of echocardiogram parameters | Day 30
  Cardiac structure and function will be measured by echocardiogram
New York Heart Association (NYHA) Functional Classification | Day 30
  NYHA Functional Classification will be determined
Results from 6-Minute Walk Test | Day 30
  Total distance walked in 6 minutes will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (48):
- United States (35):
  - Clinical Trial Site, Little Rock, Arkansas
  - Clinical Trial Site, Bakersfield, California
  - Clinical Trial Site, La Mesa, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Torrance, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Athens, Georgia
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Macon, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Merrillville, Indiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Springfield, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Jackson, Mississippi
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Camden, New Jersey
  - Clinical Trial Site, Rochester, New York
  - Clinical Trial Site, Rosedale, New York
  - Clinical Trial Site, The Bronx, New York
  - Clinical Trial Site, Williamsville, New York
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Charleston, South Carolina
  - Clinical Trial Site, Fort Worth, Texas
  - Clinical Trial Site, Plano, Texas
  - Clinical Trial Site, Falls Church, Virginia
  - Clinical Trial Site, Norfolk, Virginia
  - Clinical Trial Site, Richmond, Virginia
- Belgium (4):
  - Clinical Trial Site, Anderlecht
  - Clinical Trial Site, Brussels
  - Clinical Trial Site, Hasselt
  - Clinical Trial Site, Roeselare
- Clinical Trial Site, Blumenau, Brazil
- France (3):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Toulouse
  - Clinical Trial Site, Vandœuvre-lès-Nancy
- Spain (3):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Seville
- United Kingdom (2):
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: Undecided